CLINICAL TRIAL: NCT05188612
Title: International Survey of Acute Coronavirus Syndromes (ISACS)-COVID-19
Brief Title: International Survey of Acute Coronavirus Syndromes-COVID-19
Acronym: ISACS-COVID-19
Status: Recruiting | Type: Observational
Sponsor: University of Bologna (Other)
Collaborators: Associazione Per La Ricerca Cardiologica (Roma) (Unknown)
Responsible Party: Principal Investigator, Raffaele Bugiardini, Professor, University of Bologna
Other Study IDs: ISACS-COVID-19
Record Dates: First submitted 2022-01-08; First posted 2022-01-12 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Databases with significant genomic data (e.g., genome-wide association studies, medical sequencing, molecular diagnostic assays), are expected to be deposited as well. Likewise, physical bio-samples can be included in the ISACS-COVID-19 registry
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (10):
- Male: Non-interventional patient registry
  Interventions: Combination Product: Observational (registry)
- Female: Non-interventional patient registry
  Interventions: Combination Product: Observational (registry)
- Elderly: Non-interventional patient registry
  Interventions: Combination Product: Observational (registry)
- Hypertension: Non-interventional patient registry
  Interventions: Combination Product: Observational (registry)
- Diabetes: Non-interventional patient registry
  Interventions: Combination Product: Observational (registry)
- Dyslipidemias: Non-interventional patient registry
  Interventions: Combination Product: Observational (registry)
- Smoking: Non-interventional patient registry
  Interventions: Combination Product: Observational (registry)
- Kidney Disease: Non-interventional patient registry
  Interventions: Combination Product: Observational (registry)
- Heart Diseases: Non-interventional patient registry
  Interventions: Combination Product: Observational (registry)
- Vascular diseases: Non-interventional patient registry
  Interventions: Combination Product: Observational (registry)

INTERVENTIONS:
Combination Product: Observational (registry) — Observational (Patient Registry)

SUMMARY:
In response to the COVID-19 crisis, ISACS-TC has promoted a new registry of the existing and further centers of the same geographic areas to support clinical research to prevent, and treat the COVID-19 illness. These efforts are made possible by the generous contributions of clinical research volunteers in some of the countries participating to the prior acute coronary syndrome network.

DETAILED DESCRIPTION:
To address existing gaps in knowledge on CVD among European countries at different income levels, a collaboration of outcomes-oriented researchers from the University of Bologna partnered with Central and East European (CEE) countries researchers to conduct the International Survey of Acute Coronary Syndromes in Transitional Countries (ISACS-TC) investigating underlying threats in patients' CVD health status (NCT01218776).

In response to the COVID-19 crisis, ISACS-TC has promoted a new registry of the existing and further centers of the same geographic areas to support clinical research to prevent, and treat the COVID-19 illness. These efforts are made possible by the generous contributions of clinical research volunteers in some of the countries participating to the prior acute coronary syndrome network.

Scientific and clinical evidence is evolving on the effects of COVID-19, which can affect multiple organ systems. As, so the COVID-19 pandemic underscores the urgent need for coordination, collaboration, and information-sharing among researchers worldwide. Researchers of many disciplines have, therefore, joined the ISACS-TC investigators to build a multi-disciplinary registry investigating the impact of COVID-19.

Projects should be mainly focused on topics related to:

1. The impact of COVID-19 infection on patients who have attended any health care center (within hospital beds), and who have been discharged or have died at the time of the evaluation. The main objective of this task is to carefully characterize the clinical profile of patients infected with COVID-19 in order to develop a simple prognostic clinical score allowing rapid logistic decision making such as discharge with follow-up, referral to provisional hospitals, or admission to hospital centers with advanced equipment or specialized procedures and techniques. A secondary objective of this retrospective analysis is to evaluate the risk-adjusted influence of prior evidence-based treatments and comorbidities on patients infected with the disease.
2. The second issue relates to the long-term health consequences after COVID-19 infection. Early reports suggest residual effects of SARS-CoV-2 infection, such as fatigue, dyspnea, chest pain, cognitive disturbances, arthralgia, and decline in quality of life. However, the evidence is still scarce. Prior studies did not take into account the vast majority of patients with a mild course of the infection. As well, the definition of the post-acute COVID-19 timeline is evolving. Today we may summarize the post-acute COVID-19 syndrome into two categories:

   * subacute or ongoing symptomatic COVID-19, which includes symptoms and abnormalities present from 4-12 weeks beyond acute COVID-19;
   * chronic or post-COVID-19 syndrome, which includes symptoms and abnormalities persisting or present beyond 12 weeks of the onset of acute COVID-19 and not attributable to alternative diagnoses. Systematic study of sequelae after recovery from acute COVID-19 is needed to develop an evidence-based multidisciplinary team approach for caring for these patients, and to inform research priorities.

One trained physician will critically review the patients' reported symptoms and will assess SARS-CoV-2 IgG at each visit. In addition, wherever needed, the investigators will investigate the daily living status of survivors of COVID-19 using telephone interview questionnaires including Activity Daily Living (ADL), Self-rating Depression Scale (SDS), and New York Heart Association (NYHA) functional class.

* Sponsor: Raffaele Bugiardini (Principal Investigator; PI) - University of Bologna
* Co-PI Investigator (Clinical Research): Olivia Manfrini (University of Bologna)
* Co-PI Investigator (Translational Research): Lina Badimon (IR-Hospital de la Santa Creu i Sant Pau, UAB, Barcelona)
* Collaborator: Associazione Per La Ricerca Cardiologica, Roma

National Investigators:

Bosnia and Herzegovina: Local PI: Mirza Dilic (Clinical Center University of Sarajevo)

Croatia: Local PI: Davor Miličić (University Hospital Center Zagreb)

Other Investigators:

* Marijan Pašalić (University Hospital Center Zagreb)
* Petra Mjehović (University Hospital Center Zagreb)

Italy: Local PI: Stefano Nava (University of Bologna)

Other Investigators:

* Gaetano Caramori (University of Messina)
* Antonio David, (University of Messina)
* Giuseppe Mancuso (University of Messina)
* Maria Laura Vega Pitao (University of Bologna)
* Giulia Panzuti (University of Bologna)
* Edina Cenko (University of Bologna)
* Maria Bergami (University of Bologna)
* Marialuisa Scarpone (University of Bologna)
* Antonio Spanevello (IRCCS Maugeri)
* Fabio Angeli (IRCCS Maugeri)
* Dina Visca (IRCCS Maugeri)
* Martina Zappa (IRCCS Maugeri)
* Paolo Emilio Puddu (Associazione Per La Ricerca Cardiologica, Roma)

Macedonia: Local PI: Sasko Kedev and Marija Vavlukis (University "Ss. Cyril and Methodius")

Other Investigators:

* Lidija Poposka (University Clinic of Cardiology)
* Milena Stefanovic (University Clinic of Infectious Diseases)
* Ilir Demiri (University Clinic of Infectious Diseases) Romania: Local PI: Maria Dorobantu (Emergency Clinical Hospital of Bucharest) Other Investigators: Oana Fronea Gheorghe (Emergency Clinical Hospital of Bucharest)

Serbia: Local PI: Marija Zdravkovic (Hospital Medical Center Bezanijska kosa, Belgrade), Zorana Vasiljevic (University of Belgrade)

Other Investigators:

* Nebojsa Ladjevic, Clinic for Anesthesia, Covid Hospital Batajnica, Belgrade
* Radmilo Jankovic (Clinical Center Nis)
* Goran Loncar (Institute for Cardiovascular Diseases Dedinje)
* Ratko Lasica (Clinical Center of Serbia)
* Miodrag Petrović (Institute for Cardiovascular Diseases Sremska Kamenica, Novi Sad)
* Vlada Vukomanovic (Clinical Hospital Center Dragiša Mišković Belgrade)
* Dubravka Rajic (Clinical Center of Serbia)
* Ana Uscumlic (Clinical Center of Serbia)
* Sanja Stankovic (Clinical Center of Serbia)

Spain: Local PI: Teresa Padro (IR-Hospital de la Santa Creu i Sant Pau, UAB, Barcelona)

Other Investigators:

* Guiomar Mendieta ( CNIC, Madrid)
* Rosa Suades (IR-Hospital de la Santa Creu i Sant Pau, UAB, Barcelona)
* Gemma Vilahur (IR-Hospital de la Santa Creu i Sant Pau, UAB, Barcelona)

United Kingdom: Local PI: Charalambos Antoniades (Oxford University)

Other Investigators:

* Maria Lyasheva (University of Oxford)
* Lucy Kingham (University of Oxford)
* Christos Kotanidis (University of Oxford)
* Cheng Xie (University of Oxford)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years (male or female)
* Patients admitted to any hospital center with a confirmed diagnosis of COVID-19 infection.

Exclusion Criteria:

• Underage or not able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Confirmed diagnosis of COVID-19 infection.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Death all cause | 30-day
  Occurrence of all cause death
Death all cause | 6 month
  Occurrence of all cause death
Death all cause | 12-month
  Occurrence of all cause death

SECONDARY OUTCOMES:
Heart failure | 30 day, 6 -12 months
  Occurrence of heart failure or worsening of preexisting heart failure (According to the attending physician)
Worsening renal function | 30 day, 6 -12 months
  Occurrence of kidney disease or worsening of preexisting kidney failure (According to the attending physician)
Respiratory Insufficiency | 30 day, 6 -12 months
  Occurrence of respiratory insufficiency or worsening of preexisting respiratory insufficiency (According to the attending physician)
Pneumonia | 30 day, 6 -12 months
  Occurrence of pneumonia (According to the attending physician)
Sepsis | 30 day, 6 -12 months
  Occurrence of sepsis (According to the attending physician)
Systemic Inflammatory Response Syndrome (SIRS) | 30 day, 6 -12 months
  Occurrence of SIRS (According to the attending physician)
Thrombosis (arterial, venous) | 30 day, 6 -12 months
  Occurrence of thrombosis and thromboembolism (According to the attending physician)
Clinically relevant bleeding | 30 day, 6 -12 months
  Occurrence of clinically relevant bleeding (According to the attending physician)
Activity Daily Living status | 30 day, 6 -12 months
  (According to the attending physician)
Depression status | 30 day, 6 -12 months
  (According to the attending physician)

CONTACTS AND LOCATIONS:
Overall Officials: Olivia Manfrini, MD, Study Director — University of Bologna; Lina Badimon, PhD, Study Director — IR-Hospital de la Santa Creu i Sant Pau, UAB, Barcelona
Locations (2):
- University of Bologna, Bologna, Bologna, Italy
- IR-Hospital de la Santa Creu i Sant Pau, UAB, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bugiardini R, Nava S, Caramori G, Yoon J, Badimon L, Bergami M, Cenko E, David A, Demiri I, Dorobantu M, Fronea O, Jankovic R, Kedev S, Ladjevic N, Lasica R, Loncar G, Mancuso G, Mendieta G, Milicic D, Mjehovic P, Pasalic M, Petrovic M, Poposka L, Scarpone M, Stefanovic M, van der Schaar M, Vasiljevic Z, Vavlukis M, Vega Pittao ML, Vukomanovic V, Zdravkovic M, Manfrini O. Sex differences and disparities in cardiovascular outcomes of COVID-19. Cardiovasc Res. 2023 May 22;119(5):1190-1201. doi: 10.1093/cvr/cvad011. PMID 36651866
- [Derived] Bergami M, Manfrini O, Nava S, Caramori G, Yoon J, Badimon L, Cenko E, David A, Demiri I, Dorobantu M, Fabin N, Gheorghe-Fronea O, Jankovic R, Kedev S, Ladjevic N, Lasica R, Loncar G, Mancuso G, Mendieta G, Milicic D, Mjehovic P, Pasalic M, Petrovic M, Poposka L, Scarpone M, Stefanovic M, van der Schaar M, Vasiljevic Z, Vavlukis M, Vega Pittao ML, Vukomanovic V, Zdravkovic M, Bugiardini R. Relationship Between Azithromycin and Cardiovascular Outcomes in Unvaccinated Patients With COVID-19 and Preexisting Cardiovascular Disease. J Am Heart Assoc. 2023 Jul 18;12(14):e028939. doi: 10.1161/JAHA.122.028939. Epub 2023 Jul 14. PMID 37449568